CLINICAL TRIAL: NCT05554731
Title: Development and Application of a New Balloon Catheter for Intraairway Hemostasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020C03067
Record Dates: First submitted 2021-12-19; First posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Hemoptysis
MeSH Terms: conditions — Hemoptysis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New balloon catheter for Endotracheal hemostasis + Traditional Therapy (Experimental): 1. Haemoptysis clinic for regular haemoptysis after treatment and life safety safeguard measures;
  2. Balloon closure after informed consent (it can be blocked in emergency);
  3. CTA (can be performed as an emergency prior to balloon blockage);
  4. Artery interventional therapy (if necessary);
  5. Surgery (if needed).
  Interventions: Device: a New Balloon Catheter for Intraairway Hemostasis; Device: Traditional Therapy
- Traditional Therapy (Active Comparator): 1. Haemoptysis clinic for regular haemoptysis after treatment and life safety safeguard measures;
  2. CTA (can be performed as an emergency prior to balloon blockage);
  3. Artery interventional therapy (if necessary);
  4. Surgery (if needed).
  Interventions: Device: a New Balloon Catheter for Intraairway Hemostasis; Device: Traditional Therapy

INTERVENTIONS:
Device: a New Balloon Catheter for Intraairway Hemostasis — In the treatment group, the new balloon catheter was inserted in three steps, that is, the tracheoscope was inserted into the airway to remove the blood in the airway and find the target bronchus.The new airway hemostatic balloon catheter was directly inserted through the tracheoscopy biopsy channel, and then directly inflated and fixed after positioning.Then exit the tracheoscope directly to complete.
Device: Traditional Therapy — A six-step technique was adopted to place the traditional balloon catheter, that is, the tracheoscope was entered to find the target bronchus, the guide wire was inserted through the biopsy channel, the tracheoscope was exchanged to exit the tracheoscope, the catheter was entered through the guide wire exchange, the tracheoscope was re-entered, the catheter was positioned, inflated and fixed, and the tracheoscope was withdrawn.

SUMMARY:
Massive hemoptysis is a serious disease of respiratory system, which seriously endangers the life of patients.

There are obvious difficulties in the treatment of hemoptysis. In the traditional treatment, patients still have the risk of massive hemoptysis and suffocation, and the risk control in the treatment process cannot be ensured.

Intra - airway interventional therapy, especially the hemostatic technique of intra - airway balloon catheter, is an important means to control the risk of hemoptysis.

However, the current intraairway balloon catheter therapy technology is immature, complicated and difficult to operate, and the cost is high. There is a lack of special balloon for hemostasis, and the balloon borrowed for other purposes cannot meet the needs of hemoptysis treatment.

Therefore, it is urgent to develop a new balloon catheter for airway hemostasis, which has simple technical operation, easy to master and popularize, efficient and safe function and structure.

According to this requirement, this project designed and developed hemostatic balloon catheter with multiple functions such as self-guiding, anti-displacement, anti-leakage and detachable rear end, so as to make the treatment of massive hemoptysis more safe and effective, simpler and faster, so as to be widely applied in clinical practice.

DETAILED DESCRIPTION:
This study are aimed to investigate the safety and effectiveness of the new intraairway hemostatic balloon catheter in the treatment of massive hemoptysis, as well as the superior efficacy compared with the traditional treatment strategy of massive hemoptysis.

ELIGIBILITY:
Inclusion Criteria:

* The patients were 18-75 years, male or non-pregnant female;
* Meet the clinical definition of massive hemoptysis (blood loss ≥100ml each time or ≥500ml 24h);
* The patient/legal authorized representative understood the purpose and procedure of the test and voluntarily signed the informed consent.

Exclusion Criteria:

* Patients and their family members have no subjective treatment intention;Patients fail to cooperate or sign preoperative informed consent;
* The obvious effect of balloon catheter therapy is not ideal;
* Severe arrhythmia, acute myocardial ischemia;
* blood pressure is not effectively controlled (diastolic blood pressure ≥95mmHg or systolic blood pressure ≥150mmHg);
* Severe coagulopathy;
* Severe organ insufficiency (except respiratory insufficiency);
* Allergic to narcotic drugs;
* Pregnant women, those who are breast-feeding or trying to conceive;
* Patients who do not wish to sign informed consent;
* Patients who failed to follow up;
* Other patients deemed unsuitable for the study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Immediate intraoperative success rate | Immediately after surgery
  Immediate intraoperative success rate
Success rate of hemostasis 1 day after operation | 1 day after operation
  Success rate of hemostasis 1 day after operation
Intraoperative complication | During surgery
  Significant increase in hemoptysis requiring other emergency management or suspension of operations, asphyxia, death, new arrhythmias, persistent worsening hypoxemia.

SECONDARY OUTCOMES:
Success rate of hemostasis 3 days and 1 and 2 weeks after operation | 3 days and 1 and 2 weeks after operation
  Success rate of hemostasis 3 days and 1 and 2 weeks after operation
The bleeding time | From date of randomization until the date of second operation , assessed up to 13 months
  The bleeding time
The operation rate of balloon occlusion again | From date of randomization until the date of second operation , assessed up to 13 months
  The operation rate of balloon occlusion again
Measurement indexes of follow-up treatment measures | From date of randomization until the date of second operation , assessed up to 13 months
  Including CTA and its preparation time, rate of arterial embolization surgery and proportion of emergency surgery.
Anesthesia complications | During surgery
  Complications after anesthesia including hypotension and shock, postoperative new tracheal intubation, coma and cerebrovascular accident.
hyoxemia | From date of randomization until the date of second operation , assessed up to 13 months
  For more than 2 hours, oxygen saturation drops below 90%.
Other complications | From date of randomization until the date of second operation , assessed up to 13 months
  venous thrombosis of lower limbs
Balloon closure operation time | up to 13 months
  Compared with the traditional dilated balloon group, the operation time of balloon closure was calculated
success rate of placement | From date of randomization until death , assessed up to 13 months
  success rate of placement
time and incidence of balloon leakage | From date of randomization until the date of second operation , assessed up to 13 months
  time and incidence of balloon leakage (under the premise of two inflations per day)
incidence of balloon displacement | From date of randomization until the date of second operation , assessed up to 13 months
  incidence of balloon displacement (including the discount and distortion in the airway)
Nasal and bronchial mucosa injury | up to 13 months
  Compared with the traditional dilated balloon group, the damage of nasal and bronchial mucosa after balloon closure was observed
Rate of hemoptysis after balloon occlusion | up to 13 months
  compared with traditional balloon dilation group
Rate of re-balloon closure | up to 13 months
  compared with traditional balloon dilation group
Incomplete completion rate of balloon closure operation | up to 13 months
  compared with traditional balloon dilation group

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of wenzhou medical university, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided